CLINICAL TRIAL: NCT04543305
Title: A Phase 1, Open-Label, Multicenter, Dose-Escalation Study of PRT1419 in Patients With Relapsed/Refractory Hematologic Malignancies
Brief Title: A Study of PRT1419 in Patients With Relapsed/Refractory Hematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Prelude Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: PRT1419-01
Record Dates: First submitted 2020-09-02; First posted 2020-09-10 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-11

CONDITIONS: Multiple Myeloma; Acute Myeloid Leukemia; Non Hodgkin Lymphoma; Myelodysplastic Syndromes
MeSH Terms: conditions — Multiple Myeloma; Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin; Myelodysplastic Syndromes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PRT1419 (Experimental): PRT1419 will be administered orally
  Interventions: Drug: PRT1419

INTERVENTIONS:
Drug: PRT1419 — PRT1419 will be administered orally

SUMMARY:
This is a Phase 1 dose-escalation study of PRT1419, a myeloid cell leukemia 1 (MCL1) inhibitor, in patients with relapsed/refractory hematologic malignancies. The purpose of this study is to define the dosing schedule, maximally tolerated dose and/or estimate the optimal biological dose to be used in subsequent development of PRT1419.

DETAILED DESCRIPTION:
This is a multicenter, open-label, dose-escalation Phase 1 study of PRT1419, a MCL1 inhibitor, evaluating patients in two cohorts as part of a 28-day treatment cycle in adult patients with multiple myeloma (MM), non-Hodgkin's lymphoma (NHL), acute myeloid leukemia (AML), chronic myelomonocytic leukemia (CMML), high-risk myelodysplastic syndrome (MDS) or MDS/myeloproliferative neoplasm (MPN) overlap syndrome. Cohort A will evaluate PRT1419 administered as monotherapy in patients with either AML, CMML and/or high-risk MDS or MDS/MPN overlap. Cohort B will evaluate PRT1419 administered as monotherapy in patients with NHL or MM. The study will employ a "3+3" dose escalation design. The dose may be escalated until a dose limiting toxicity is identified.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* Adequate organ function (bone marrow, hepatic, renal, cardiovascular)
* Left ventricular ejection fraction of ≥50%
* Female patients of childbearing potential must have a negative pregnancy test within 7 days of the start of treatment and must agree to use a highly effective method of contraception during the trial
* Patients must have recovered from the effects of any prior cancer related therapy, radiotherapy or surgery (toxicity ≤ Grade 1)
* All patients on prior investigational agents must wait at least 5 half-lives of the agent in question, or 14 days, whichever is longer before study entry
* AML patients only: Pathologically confirmed diagnosis of AML as defined by the WHO Classification and patients with targeted mutations must have been treated with appropriate therapy for their disease

  * White blood cell count < 25 x 10^9/L. Hydrea or leukapheresis are permitted to meet this criterion.
* CMML patients only: intermediate-2 or high risk per CMML-specific prognostic scoring system (CPSS) or clinical/molecular CPSS (CPSS-mol) criteria. Must have failed prior therapy with a hypomethylating agent.
* MDS patients only: Intermediate, high, or very high risk by International Prognostic Scoring System-Revised [IPSS-R] criteria that is relapsed or refractory to approved therapies or MDS/MPN Overlap Syndrome (displaying both fibrosis and dysplastic features).
* NHL patients only: Histologically or cytologically confirmed NHL, including B- and T-cell lymphomas that is relapsed or refractory or intolerant to approved therapies. Must have one lesion that can be measured for response
* MM patients only: Measurable disease defined by one or more of the following: Serum M-protein ≥ 0.5 g/dL, Urine M-protein ≥ 200 mg/24 hours, Serum Free Light Chain (sFLC) > 10 mg/dL with normal serum FLC ratio. Presence of soft tissue plasmacytoma confirmed by imaging
* NHL and MM patients only: must have the following lab values within 14 days prior to study Day 1:

  * ANC ≥1.0 x 10^3 μL
  * Platelet count ≥50,000 μL

Exclusion Criteria:

* Known hypersensitivity to any of the components of PRT1419
* Female patients who are pregnant or lactating
* Mean QTcF interval of >480 msec
* History of heart failure, additional risk factors for arryhthmias or requiring concomitant medications that prolong the QT/QTc interval
* Hematopoietic stem-cell transplant < 90 days or have GVHD Grade >1 at study entry
* Uncontrolled intercurrent illnesses
* Treatment with strong inhibitors of CYP2C8 and/or P-glycoprotein for which there are no therapeutic substitutions
* Inflammatory disorders of the gastrointestinal tract, or subjects with GI malabsorption
* HIV positive; known active hepatitis B or C
* Prior exposure to an MCL1 inhibitor
* History of another malignancy except:

  * Malignancy treated with curative intent with no known active disease for >2 years at study entry
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
  * Other concurrent low-grade malignancies (i.e chronic lymphocytic leukemia (Rai 0)) may be considered after consultation with Sponsor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2022-03-21 (Actual); Study Completion 2022-03-21 (Actual)

PRIMARY OUTCOMES:
To describe dose limiting toxicities (DLT) of PRT1419 | Baseline through Day 28
  Dose limiting toxicities will be evaluated through the first cycle
To determine the maximally tolerated dose (MTD) and/or optimal biological dose (OBD) | Baseline through approximately 2 years
  The MTD and/or OBD will be established for further investigation in participants with multiple myeloma, Non-Hodgkin's Lymphoma, acute myeloid leukemia and myelodysplastic syndrome
To determine the recommended phase 2 dose (RP2D) and schedule of PRT1419 | Baseline through approximately 2 years
  The RP2D will be established for further investigation in participants with multiple myeloma, Non-Hodgkin's Lymphoma, acute myeloid leukemia and myelodysplastic syndrome

SECONDARY OUTCOMES:
To describe the adverse event profile and tolerability of PRT1419 | Baseline through approximately 2 years
  Adverse events as characterized by type, frequency, severity, timing, seriousness and relationship to study therapy
To describe the pharmacokinetic profile of PRT1419 | Baseline through approximately 2 years
  PRT1419 pharmacokinetics will be calculated including the maximum observed plasma concentration
To describe any anti-tumor activity of PRT1419 | Baseline through approximately 2 years
  Anti-tumor activity of PRT1419 will be based on the measurement of objective responses

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Florida Cancer Specialists, Lake Mary, Florida
  - Florida Cancer Specialists, Sarasota, Florida
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - The University of Texas MD Anderson Cancer Center, Houston, Texas